CLINICAL TRIAL: NCT03734744
Title: A Pilot Study Evaluating Single, High-dose Pharmacokinetics/Pharmacodynamics of Vitamin D3 in CF
Brief Title: PK/PD of Vitamin D3 in Adults With CF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical research currently on hold
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Paul Beringer, Professor of Clinical Pharmacy, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-18-00737
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Vitamin D Deficiency; Cystic Fibrosis
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Vitamin D Deficiency; Cystic Fibrosis | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults with Cystic Fibrosis (Experimental): CF adults with vitamin D insufficiency or deficiency will receive 300,000-600,000 IU vitamin D3 (cholecalciferol)
  Interventions: Dietary Supplement: Vitamin D3
- Non-CF Controls with Low vitamin D (Experimental): Non-CF controls with vitamin D insufficiency or deficiency will receive 300,000-600,000 IU vitamin D3 (cholecalciferol)
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D is a fat-soluble vitamin that plays an important role in immune modulation in addition to its classical roles in regulation of calcium homeostasis and bone health
  Other Names: Cholecalciferol

SUMMARY:
Despite the extensive literature on adverse clinical outcomes associated with vitamin D deficiency, there are currently no proven treatment strategy that effectively achieves and maintains optimal serum vitamin D status in cystic fibrosis (CF) patients. For the treatment of vitamin D deficiency, CF Foundation currently recommends 2,000 IU daily. However, because achieving adequate serum 25(OH)D levels is a challenge in CF, higher doses of vitamin D may be necessary to reach and maintain vitamin D sufficiency. Poor oral bioavailability of ergocalciferol has been demonstrated in CF patients, which may potentially also be an issue with cholecalciferol. In order to optimize the treatment of vitamin D deficiency in CF, the kinetic disposition must be well understood. However, there are very few data currently available describing the kinetics of both vitamin D and 25-hydroxyvitamin D, and to the investigator's knowledge, no studies have yet characterized the pharmacokinetic disposition of vitamin D and its metabolites in cystic fibrosis. Addressing this issue is crucial in effectively and safely correcting vitamin D deficiency in CF.

DETAILED DESCRIPTION:
Clinically stable CF patients with a history of pancreatic insufficiency (n=6) and matching non-CF subjects (n=6) will be recruited in this study. All subjects will be pre-screened for 25(OH)D status to include those with 25(OH)D levels below 30 ng/mL. The subjects will receive a single oral dose (300,000 - 600,000 IU) of vitamin D3, and the dose will be based on study participant's baseline 25-hydroxyvitamin D3 level. For CF patients, the dose will be administered with food and pancreatic enzyme supplement. This dose was chosen as previous studies in pediatric CF patients demonstrated that a large single dose of up to 600,000 IU vitamin D3 raised and maintained sufficient 25(OH)D concentrations without any signs of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* For CF, diagnosis of CF based on positive sweat chloride or known CF mutation
* For CF, Patients with pancreatic insufficiency
* Age ≥ 18 years
* Serum 25(OH)D concentrations below 30 ng/mL (75 nmol/L)

Exclusion Criteria:

* Pregnancy
* History of lung transplant,
* Severe anemia (hemoglobin concentration < 7 g/dL),
* Liver disease (AST/ALT > 3x ULN), kidney disease (GFR ≤ 40 mL/min), or granulomatous conditions
* Patients taking steroids, cholesterol-lowering drug (cholestyramine), weight-loss drugs (orlistat) , statins, anti-tuberculosis drugs (rifampin and isoniazid), phenobarbital, phenytoin, carbamazepine, immunosuppressants (cyclosporine, tacrolimus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentrations (Cmax) | 10 weeks
Time taken to reach the maximum concentration (Tmax) | 10 weeks
Area under the plasma concentration versus time curve (AUC) | 10 weeks

SECONDARY OUTCOMES:
Levels of serum inflammatory biomarkers | 10 weeks
  Changes in IL-6, IL-8, TNF-α, IL-1β, C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Beringer, Pharm.D., Principal Investigator — University of Southern California
Locations (1):
- Keck Hospital of University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thacher TD, Clarke BL. Vitamin D insufficiency. Mayo Clin Proc. 2011 Jan;86(1):50-60. doi: 10.4065/mcp.2010.0567. PMID 21193656
- [Background] Tangpricha V, Kelly A, Stephenson A, Maguiness K, Enders J, Robinson KA, Marshall BC, Borowitz D; Cystic Fibrosis Foundation Vitamin D Evidence-Based Review Committee. An update on the screening, diagnosis, management, and treatment of vitamin D deficiency in individuals with cystic fibrosis: evidence-based recommendations from the Cystic Fibrosis Foundation. J Clin Endocrinol Metab. 2012 Apr;97(4):1082-93. doi: 10.1210/jc.2011-3050. Epub 2012 Mar 7. PMID 22399505
- [Background] Shepherd D, Belessis Y, Katz T, Morton J, Field P, Jaffe A. Single high-dose oral vitamin D3 (stoss) therapy--a solution to vitamin D deficiency in children with cystic fibrosis? J Cyst Fibros. 2013 Mar;12(2):177-82. doi: 10.1016/j.jcf.2012.08.007. Epub 2012 Sep 19. PMID 22998937
- [Background] Grossmann RE, Zughaier SM, Kumari M, Seydafkan S, Lyles RH, Liu S, Sueblinvong V, Schechter MS, Stecenko AA, Ziegler TR, Tangpricha V. Pilot study of vitamin D supplementation in adults with cystic fibrosis pulmonary exacerbation: A randomized, controlled trial. Dermatoendocrinol. 2012 Apr 1;4(2):191-7. doi: 10.4161/derm.20332. PMID 22928076
- [Background] Lark RK, Lester GE, Ontjes DA, Blackwood AD, Hollis BW, Hensler MM, Aris RM. Diminished and erratic absorption of ergocalciferol in adult cystic fibrosis patients. Am J Clin Nutr. 2001 Mar;73(3):602-6. doi: 10.1093/ajcn/73.3.602. PMID 11237938

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03734744/Prot_SAP_000.pdf